CLINICAL TRIAL: NCT02601144
Title: Double-Blind Trial of Variable Frequency Stimulation for Freezing of Gait in Parkinson's Disease
Brief Title: Variable Frequency Stimulation of Subthalamic Nucleus for Freezing of Gait in Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: PINS-014
Record Dates: First submitted 2015-10-12; First posted 2015-11-10 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Parkinson's Disease
Keywords: DBS; VFS; FOG
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- VFS (Experimental): variable frequency deep brain stimulation (VFS)
  Interventions: Device: Deep Brain Stimulation
- HFS (Active Comparator): high frequency deep brain stimulation (HFS)
  Interventions: Device: Deep Brain Stimulation
- LFS (Active Comparator): low frequency deep brain stimulation (LFS)
  Interventions: Device: Deep Brain Stimulation
- DBS off (No Intervention): deep brain stimulation off

INTERVENTIONS:
Device: Deep Brain Stimulation — Deep Brain Stimulation
  Arms: HFS; LFS; VFS

SUMMARY:
This is the first study on the effect of the variable frequency stimulation (VFS) on Freezing of gait (FOG) in Parkinson's disease (PD) patients with STN DBS. FOG has responded poorly to High frequency stimulation (HFS) but can be alleviated by relatively VFS. This study would have significant clinical implications in the management of Freezing of gait (FOG) in these PD patients with subthalamic nucleus (STN) DBS. The investigators hypothesize that VFS could have better effect on FOG than HFS and low frequency stimulation (LFS).

DETAILED DESCRIPTION:
HFS of STN provides consistent, long-term improvement of the cardinal motor signs of PD, such as bradykinesia, tremor and rigidity. FOG has responded poorly to HFS and tends to continue to deteriorate over time, but this can be alleviated by relatively LFS. Evidence has indicated that LFS-STN can improve axial signs in some but not all PD patients, but most of them experienced loss of efficacy in the short term. Then comes to the little improvement or even worse of tremor, rigidity and bradykinesia, which consists of the three main symptoms of Parkinson's disease. Thus even if axial problems could be solved by LFS in a long way, it could also be hard to tolerate by those patients. The effect of VFS on FOG will be studied. The investigators hypothesize that VFS could have better effect on Freezing of gait than HFS and LFS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were receiving bilateral STN stimulation for more than six months.
2. They were optimized on conventional HFS for control of tremors, rigidity and bradykinesia yet complained of freezing of gait.
3. Subjects had an ability to walk at least 10 meters independently during ON DBS condition.

Exclusion criteria:

1. gait disorders perceived by patients as a direct consequence of STN stimulation and not the primary disease.
2. any change in the HFS DBS settings, three months prior to participation in the study.
3. complete inability to walk despite assistance while DBS ON.
4. Subjects responding to reprogramming of chronic DBS settings (report improvement of freezing).
5. Subjects could not tolerate prolonged OFF medication condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) task | The outcome of TUG task at 12 months follow-up.
  variable frequency stimulation (VFS) setting compared to high frequency stimulation (HFS) and low frequency stimulation (LFS)
the number of freezing episodes for TUG task | The outcome of TUG task at 12 months follow-up.
  variable frequency stimulation (VFS) setting compared to high frequency stimulation (HFS) and low frequency stimulation (LFS)

SECONDARY OUTCOMES:
UPDRS III scores | Outcome of VFS at 6、12 months with reference to baseline HFS
Gait and Falls Questionnaire (GFQ) scores | Outcome of VFS at 6、12 months with reference to baseline HFS
the39-item Parkinson's Disease Questionnaire (PDQ-39) scores | Outcome of VFS at 6、12 months with reference to baseline HFS
the Freezing of Gait Questionnaire (FOG-Q) scores | Outcome of VFS at 6 、12months with reference to baseline HFS
Number of adverse events (AE's) | Change from Baseline to 6、12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Luming Li, Ph.D, Study Chair — Tsinghua University; Michael Okun, MD., Study Chair — University of Florida
Locations (2):
- China (2):
  - Tsinghua University Yuquan Hospital, Beijing, Beijing Municipality
  - Beijing Tian Tan Hospital,Capital Medical University, Beijing, Beijing Municipality